CLINICAL TRIAL: NCT03029949
Title: Acceptance and Commitment Therapy With Vestibular Rehabilitation for Chronic Dizziness: a Randomized Controlled Trial
Brief Title: Acceptance and Commitment Therapy With Vestibular Rehabilitation for Chronic Dizziness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nagoya City University (Other)
Responsible Party: Principal Investigator, Masaki Kondo, MD, PhD, Nagoya City University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Chronic Dizziness
Keywords: chronic dizziness; persistent postural-perceptual dizziness; acceptance and commitment therapy; behavior therapy; vestibular rehabilitation

STUDY DESIGN:
Masking Description: Statisticians are blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT with VR (Experimental): acceptance and commitment therapy with vestibular rehabilitation in addition to clinical management
  Interventions: Behavioral: ACT with VR; Other: clinical management
- Self-treatment VR (Active Comparator): self-treatment vestibular rehabilitation in addition to clinical management
  Interventions: Behavioral: self-treatment VR; Other: clinical management

INTERVENTIONS:
Behavioral: ACT with VR — 6 weekly 120-minute group sessions of acceptance and commitment therapy with vestibular rehabilitation, and brief (approximately 15 minute) individual follow-up sessions at 1 and 3 months after the group treatment
  Arms: ACT with VR
Behavioral: self-treatment VR — booklet written on vestibular rehabilitation for self-treatment
  Arms: Self-treatment VR
Other: clinical management — clinical management and pharmacotherapy as usual for chronic dizziness

SUMMARY:
The purpose of this study is to examine the effectiveness of group acceptance and commitment therapy with vestibular rehabilitation for chronic dizziness, in comparison with self-treatment vestibular rehabilitation in addition to clinical management.

DETAILED DESCRIPTION:
The purpose of this study is to examine whether group acceptance and commitment therapy combined with vestibular rehabilitation in addition to clinical management for patients with persistent postural-perceptual dizziness is more effective than treatment-as-usual(TAU), which is self-treatment vestibular rehabilitation in addition to clinical management.

ELIGIBILITY:
Inclusion Criteria:

* Persistent postural-perceptual dizziness (diagnosed by the diagnostic guideline of ICD-11 beta version at Dec. 2016)
* Existing handicap due to dizziness (DHI equal to or more than 16)
* Written consent

Exclusion Criteria:

* Vertigo/dizziness/unsteadiness by organic brain diseases, diagnosed by neuro-otologist
* Vertigo/dizziness/unsteadiness explained by only organic cause or drug, diagnosed by neuro-otologist
* Physical status inappropriate for psychotherapy or vestibular rehabilitation
* Current psychiatric disorder other than anxiety disorders, somatic symptom disorder, or illness anxiety disorder (DSM-5), diagnosed by psychiatrist
* History of schizophrenia or bipolar disorder diagnosed by psychiatrist
* Increased risk of suicide or self-harm diagnosed by psychiatrist
* Started or increased SSRI/Venlafaxine within 1 month before treatment
* Any cognitive behavioral therapy or vestibular rehabilitation except this study
* Otological surgery or device therapy for dizziness
* Insufficient understanding of the Japanese language

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Handicap due to dizziness | Post-treatment and 1, 3, and 6 months after treatment (The time point of primary interest is 3 months after treatment.)
  The total score of Dizziness Handicap Inventory (DHI) (The DHI scores range from 0 to 100 points. The higher the score, the greater the handicap.)

SECONDARY OUTCOMES:
Response | Post-treatment and 1, 3, and 6 months after treatment
  Decrease in the total score of DHI equal to or more than 11
Remission | Post-treatment and 1, 3, and 6 months after treatment
  The total score of DHI equal to or less than 14
Frequency of dizziness-related symptoms | Post-treatment and 1, 3, and 6 months after treatment
  The total score of Vertigo Symptom Scale-short form (VSS-sf) (The VSS-sf scores range from 0 to 60 points. The higher the score, the worse.)
Anxiety | Post-treatment and 1, 3, and 6 months after treatment
  The anxiety subscale score of Hospital Anxiety and Depression Scale (HADS) (The HADS-anxiety scores range from 0 to 21 points. The higher the score, the worse.)
Depression | Post-treatment and 1, 3, and 6 months after treatment
  The depression subscale score of HADS (The HADS-depression scores range from 0 to 21 points. The higher the score, the worse.)
Recovery process | Post-treatment and 1, 3, and 6 months after treatment
  The total score of Recovery Assessment Scale (RAS) (The RAS scores range from 24 to 120 points. The higher the score, the better.)
Health-related quality of life | Post-treatment and 1, 3, and 6 months after treatment
  The score of EuroQOL 5 dimensions 5-level (EQ-5D-5L) (The EQ-5D-5L scores range from 0 to 1. The higher the score, the better.)
Valued living (progress, obstruction) | Post-treatment and 1, 3, and 6 months after treatment
  The each subscale score of Valuing Questionnaire (VQ) (The scores for both VQ-progress and VQ-obstruction range from 0 to 30. The higher the VQ-progress score, the better; the higher the VQ-obstruction score, the worse.)
Cognitive fusion | Post-treatment and 1, 3, and 6 months after treatment
  The total score of Cognitive Fusion Questionnaire (CFQ) (The CFQ scores range from 7 to 49 points. The higher the score, the worse.)
Somatic symptom burden | Post-treatment and 1, 3, and 6 months after treatment
  The total score of Somatic Symptom Scale-8 (SSS-8) (The SSS-8 scores range from 0 to 32. The higher the score, the worse.)

CONTACTS AND LOCATIONS:
Overall Officials: Masaki Kondo, MD, PhD, Principal Investigator — Nagoya City University
Locations (1):
- Nagoya City University, Nagoya, Aichi-ken, Japan

IPD SHARING:
Plan to Share IPD: Undecided